CLINICAL TRIAL: NCT05514132
Title: A Phase I, Multi-centre, Open-label, Dose Exploration Study to Assess the Safety and Tolerability of Ceralasertib in Combination With Durvalumab in Chinese Patients With Advanced Solid Tumours
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Ceralasertib in Combination With Durvalumab in Chinese Patients With Advanced Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5330C00017
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumours
Keywords: Phase 1; Safety; Tolerability; Pharmacokinetics; Advanced solid tumours
MeSH Terms: interventions — ceralasertib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ceralasertib in Combination with Durvalumab (Experimental): This is a sequential group treatment/dose-escalation study with 2 cohorts with no masking.
  Interventions: Drug: Ceralasertib; Drug: Durvalumab

INTERVENTIONS:
Drug: Ceralasertib — Ceralasertib (AZD6738) is a potent, selective inhibitor of the serine/threonine-specific protein kinase, ATR, with good selectivity against other phosphatidylinositol 3-kinase-related kinase family members.
  Other Names: Ceralasertib taken orally
Drug: Durvalumab — Durvalumab is a human mAb of the immunoglobulin G 1 kappa subclass that blocks the interaction of PD-L1 (but not PD-L2) with PD-1 on T cells and CD80 (B7.1) on immune cells.
  Other Names: Durvalumab Infusion

SUMMARY:
This is a Phase 1, open-label study of ceralasertib given in combination with durvalumab in Chinese participants with advanced solid tumours. In each cohort, a monotherapy lead-in period (Cycle 0, duration of 7 or 14 days), prior to dosing with durvalumab, is added to investigate the PK profile and safety/tolerability of ceralasertib in Chinese participants.

This study is designed to investigate and characterise preliminary safety, tolerability, and PK of ceralasertib in DLT-evaluable Chinese participants

DETAILED DESCRIPTION:
<Objectives>

Primary Objective:

To assess the safety and tolerability of ceralasertib in combination with durvalumab in Chinese patients with advanced solid tumours refractory/resistant to prior SoC therapy or for which no appropriate SoC therapy exists.

Secondary Objective:

To characterise the PK profile of ceralasertib after single- and multiple-doses administration. To characterise the anti-tumour activity and efficacy of ceralasertib in combination with durvalumab in Chinese patients .

<Overall design> This is a Phase 1, open-label study of ceralasertib given in combination with durvalumab in Chinese patients with advanced solid tumours.Results from this study will provide dose rationale for future investigations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. At least 18 years of age at the time of signing the ICF.
3. Histological or cytological confirmation advanced solid tumour with refractory/resistance to a prior line of anti-PD-1/PD-L1-containing therapy (received as monotherapy or in combination) or for which no SoC exists.
4. Ability to swallow oral medication intact and retain it.
5. ECOG/WHO performance status of 0 to 1.
6. Must have a life expectancy of at least 12 weeks.
7. Participant must have had a treatment-free interval of ≥ 3 weeks from any prior therapy before the first dose of study treatment.
8. Body weight > 35 kg and no cancer-associated cachexia (eg, CTCAE Grade 2 or worse weight loss over the 3 months prior to the Screening Visit).
9. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Inadequate bone marrow reserve or organ function
2. As judged by the investigator, any evidence of uncontrolled intercurrent illness, that in the investigator's opinion makes it undesirable for the participant to participate in the study.
3. Spinal cord compression, leptomeningeal disease, or brain metastases, unless asymptomatic, treated, stable, and not requiring continuous corticosteroids
4. As judged by the investigator, any active disease or condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy
5. History of another primary malignancy.
6. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, active bleeding diatheses, renal transplant, or active infection including any patient known to have hepatitis B, hepatitis C, and HIV.
7. Known history of HIV infection.
8. Active cardiacvascular disease be consider as clinical significant.
9. Active or prior documented autoimmune or inflammatory disorders
10. Prior exposure to a CHK1 or ATR inhibitor.
11. As judged by the investigator, any unresolved treatment-related toxicities from previous anti-cancer therapy of CTCAE v5.0 Grade ≥ 2
12. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment.
13. Participants must not have experienced a toxicity that led to permanent discontinuation of prior anti-PD-1 or anti-PD-L1 immunotherapy.
14. Participants must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged
15. Participants with a known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
16. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
17. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
18. Previous enrolment in the present study.
19. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity, as defined in the protocol. | From the first dose of study treatment Up to and including the end of cycle 1(each cycle is 28 days) .
  Dose-limiting toxicity as described in the protocol that is not related to disease progression, intercurrent illness or concomitant medications and that, despite optional therapeutic intervention, meets protocol-defined criteria.
Safety and tolerability in terms of adverse events | From the first dose of study treatment until 28 days after the last dose.
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters

SECONDARY OUTCOMES:
Plasma ceralasertib concentration(Cmax) | Cycle 0 Day1 to Day7, Cycle1 Day1 and Cycle 1 Day 7 or Day 8. At the end of Cycle1(each cycle is 28 days)
  Observed PK parameters of ceralasertib
Area under the plasma concentration versus time curve(AUC) | Cycle 0 Day1 to Day7, Cycle1 Day1 and Cycle1 Day7 or Day8. At the end of Cycle1(each cycle is 28 days)
  Observed PK parameters of ceralasertib.
Overall response rate | At screening and Every 8 weeks ±1 week relative to the start of therapy (Cycle 1 Day 1, each cycle is 28days) until objective disease progression as defined by RECIST version 1.1
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Duration of Response | At screening and Every 8 weeks ±1 week relative to the start of therapy (Cycle 1 Day 1, each cycle is 28 days) until objective disease progression as defined by RECIST version 1.1
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Percentage Change in Tumour Size | At screening and Every 8 weeks ±1 week relative to the start of therapy (Cycle 1 Day 1, each cycle is 28 days) until objective disease progression as defined by RECIST version 1.1
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1
Progression Free Survival | From start of treatment until the date of objective disease progression or death. (approximately 6 months).
  Antitumor activity by evaluation of tumor response assessments using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, PHD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Research Site, Beijing
  - Research Site, Shandong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluatedas per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level datain an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home